CLINICAL TRIAL: NCT06234904
Title: An Open-label, Multi-center, Phase I Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of IBR733 Cell Injection in Acute Myeloid Leukemia
Brief Title: Study of IBR733 Cell Injection in Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imbioray (Hangzhou) Biomedicine Co., Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IBR733-101
Record Dates: First submitted 2024-01-21; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; R/R AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBR733 Cell Injection (Experimental)
  Interventions: Biological: IBR733 Cell Injection

INTERVENTIONS:
Biological: IBR733 Cell Injection — The minimum initial dose is 5.0×10^9 cells and then escalate to 7.5×10^9 cells and 10.0×10^9 cells. Every 21 days is one cycle, and intravenous infusion is performed on day 1 and day 8 of each cycle.

SUMMARY:
This is an open-label clinical study: phase Ia is the dose-escalation part, and phase Ib is the dose-expansion part. The phase Ia study is to evaluate the safety, tolerability, recommended phase II dose, pharmacokinetics, immunogenicity and preliminary efficacy of IBR733 cell injection in relapsed/refractory acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Phase Ia is the dose escalation part which adopts the "3+3" dose escalation design protocol. The dose is respectively 5.0×10^9 cells, 7.5×10^9 cells and 10.0×10^9 cells. 3-6 subjects will be enrolled at every dose level. Subjects who have signed the Informed Consent Form (ICF) will be reviewed for inclusion/exclusion criteria (this process is called "screening"), and eligible subjects will be treated with IBR733 cell injection after lymphodepletion therapy. The administration of IBR733 cell injection is performed on day 1 and day 8 of each cycle (21 days). The first and second subjects in the same group shall be enrolled at an interval of at least 21 days, for the purpose of ensuring their safety.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects volunteer to participate in this clinical study, are fully aware of the study and have signed the Informed Consent Form (ICF). Subjects are willing to follow and able to complete all trial procedures.
2. Age: 18-74 (both inclusive), female or male.
3. Patients with AML (including secondary AML) diagnosed according to the WHO 2022 criteria.
4. Patients with AML who meet one of the following criteria: (1) Relapsed AML: reoccurrence of leukemia cells in peripheral blood or ≥5% blasts in bone marrow after complete remission (excluding other causes such as bone marrow regrowth after consolidation chemotherapy); (2) Refractory AML: treatment-naive patients who failed to respond to 2 courses of standard treatment; The patients relapsed within 12 months after consolidated intensive treatment; Patients who relapsed after 12 months but failed to respond to conventional chemotherapy (only once); Patients who are relapsed twice; (3) Patients received up to 3 additional cycles of chemotherapy or targeted therapy after the diagnosis of relapsed/refractory AML.
5. Eastern Cooperative Oncology Group (ECOG) score ≤2.
6. Subjects of reproductive age and their partners should agree to have no family planning and to use effective contraceptive methods for 6 months from signing the ICF until the last dose of the study drug is administered.
7. Expected survival time ≥3 months.

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Chronic myeloid leukemia with myeloid blast crisis.
3. Clinically symptomatic central nervous system involvement (no need for lumbar puncture).
4. Subjects who have undergone an allogeneic hematopoietic stem cell transplantation or other organ transplantation.
5. Subjects who have undergone autologous hematopoietic stem cell transplantation less than 3 months before the first dose of treatment.
6. Subjects who have received cell immunotherapy such as chimeric antigen receptor-modified T cells (CAR-T), chimeric antigen receptor-natural killer cells (CAR-NK), and T cell receptor gene-modified T cells (TCR-T).
7. Subjects who have received systemic antitumor therapy (except hydroxyurea) within 2 weeks before the first dose of study drug, including chemotherapy, immunotherapy, etc..
8. Subjects who have had other malignant tumors within 3 years before inclusion, except for any type of carcinoma in situ that has been cured in the past and cured skin basal cell carcinoma or skin squamous cell carcinoma.
9. The absolute peripheral blood blast count (ABC) > 40.0×10^9/L (ABC= total white blood cell count × blast %). The total white blood cell count can be controlled with hydroxyurea, but it must be stopped three days before the first dose of study drug or lymphodepletion.
10. Organ function: (1) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)>3 times upper limit of normal (ULN); If AST was elevated due to leukemia but liver function was normal (e.g., normal ALT, alkaline phosphatase, and direct/indirect bilirubin measurements), participants could be enrolled after investigator consent was obtained; (2) Serum total bilirubin >2.5×ULN (not applicable to patients with Gilbert's syndrome); (3) Creatinine clearance <45mL/min (estimated by Cockcroft-Gault formula) or creatinine >2×ULN; (4) Activated partial thromboplastin time >1.5×ULN or international normalized ratio >1.5×ULN.
11. Subjects whose cardiac function and disease meet one of the following conditions within 6 months before the first administration: (1) Any risk factors that increase QTcF (Fridericia formula) interval prolongation, such as uncorrectable hypokalemia, hereditary long QT syndrome, and use of drugs that prolong the QTcF interval; (2) New York Heart Association (NYHA) classification ≥Grade 3; (3) Unstable angina pectoris, and myocardial infarction; (4) Left ventricular ejection fraction <50% in resting state; (5) Clinically significant pericardial effusion determined by echocardiography.
12. Subjects who have a history of autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.) that require systemic immunosuppressive/systemic disease modulating drugs within 2 years before the first administration.
13. Active hepatitis B (e.g., DNA copy number > 1000 cps/mL if only hepatitis B surface antigen is positive), active hepatitis C virus infection (anti-hepatitis C antibody positive and HCV RNA positive), or human immunodeficiency virus antibody positive.
14. Women who are pregnant or lactating.
15. Subjects who have received major surgery (for the definition of major surgery, refer to the Level 3 and 4 surgeries specified in the Administrative Measures for the Clinical Application of Medical Technology) within 28 days before the first administration.
16. Subjects who have a history of alcohol, drug use or drug abuse in the past year;
17. Subjects who have participated in other clinical trials and received any unmarketed investigational drug or treatment within 4 weeks prior to first use of the study drug.
18. Subjects who are known to be allergic to the main components of the study drug.
19. Subjects who have other severe, acute, or chronic diseases or laboratory abnormalities that may increase the risk of participating in the study and receiving the study drug, or may interfere with the interpretation of study results.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | From day1 to day 21
  To evaluate the safety, tolerability, and determine the RP2D of IBR733 cell injection
The incidence and severity of adverse events (AEs) | From day 1 to day 30 after the last dose
  To evaluate the safety of IBR733 cell injection

SECONDARY OUTCOMES:
Complete remission rate (CRR) | From day 1 up to 6 weeks
  The rate of subjects who achieved complete remission (CR) among all subjects
Composite complete remission rate | From day 1 up to 6 weeks
  The rate of subjects achieving complete remission (CR) and complete remission with incomplete hematologic recovery (CRi) or complete remission with partial hematologic recovery (CRh) among all subjects
Objective remission rate (ORR) | From day 1 up to 6 weeks
  The rate of subjects achieving CR, CRi, morphologic leukemia-free state(MLFS), and partial remission(PR) among all subjects
Duration of remission (DOR) | From day 1 up to 3 months
  Time from the subject's first assessment of the onset of remission to the first assessment of disease recurrence or progression or death from any cause
Overall survival (OS) | From day 1 up to 3 months
  Time from the start of treatment to death from any cause
The number of IBR733 cells | From day1 to day 21
  Blood samples will be collected at specified time points to detect the number of IBR733 cells in peripheral blood
Anti-drug antibodies | From day1 up to 6 weeks
  Blood samples will be collected at specified time points to detect anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China